CLINICAL TRIAL: NCT00563199
Title: A Randomized Controlled Trial of a Nurse Delivered Stage-matched Smoking Cessation Intervention to Promote Heart Health of Cardiac Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Authority, Hong Kong (Other Government)
Collaborators: Research Grants Council, Hong Kong (Other)
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: NTWC/CREC/325/04; HARECCTR0500022; HKU 7224/01M
Record Dates: First submitted 2007-11-21; First posted 2007-11-26 (Estimated); Last update posted 2011-06-16 (Estimated); Status verified 2011-06

CONDITIONS: Smoking Cessation; Smoking
Keywords: smoking cessation; smoking behaviors
MeSH Terms: conditions — Smoking Cessation; Smoking

INTERVENTIONS:
Behavioral: nurse-delivered stage-matched smoking cessation counseling

SUMMARY:
This study is a randomized controlled trial designed to evaluate the effectiveness of a nurse delivered stage-matched intervention to cardiac patients for cessation of tobacco use. Review of literature shows that there is a clear lack of empirical evidence on (1) using nurses to deliver stage-matched smoking cessation interventions, and (2) the effectiveness of such intervention for cardiac patients in Chinese populations. The ultimate goal of the intervention achieve a higher quit rate in the intervention group than in the controls. In addition, the change in the patient's smoking behaviour such as reduction of the number of cigarettes smoked, and progression to a higher stage of readiness to quit, will also be measured. This study is the first step to address the urgently needed data for (1) promoting the delivery of nurse-run stage-matched smoking cessation interventions to help patients stop smoking, (2) developing smoking cessation policy and programmes in the hospitals and for the health care system, and (3) contributing an evidence-based approach to orientate clinical services towards prevention, so as to reduce premature deaths and the enormous disease burden of our society.

ELIGIBILITY:
Inclusion Criteria:

* Patient who is admitted to the participating centres and is a current smoker who has smoked daily in the past 7 days prior to hospitalization.
* Patient speaks and reads Cantonese/Chinese

Exclusion Criteria:

* Patient who is clinically too ill and not suitable to complete questionnaire and/or receive intervention.
* Patient who does not speak or read Chinese

Sex: All
Age Groups: Child, Adult, Older Adult
Enrollment: 1824 (Estimated)
Dates: Start 2002-03; Study Completion 2005-12 (Actual)

PRIMARY OUTCOMES:
Quitting--to achieve higher quit rate in the cardiac patients (coronary artery disease) who are smokers | continuous abstinence for one month at the time of 3, 6 and 12 month follow up

SECONDARY OUTCOMES:
Reduction of the number of cigarettes smoked | at the time of 3, 6 and 12 month follow up
Progression to a higher stage of readiness to quit | at the time of 3, 6 and 12 month follow up

CONTACTS AND LOCATIONS:
Overall Officials: Sophia SC Chan, Dr, Principal Investigator — Department of Nursing Studies, The University of Hong Kong
Locations (10):
- China (10):
  - Caritas Medical Centre, Hong Kong
  - Pamela Youde Nethersole Eastern Hospital, Hong Kong
  - Princess Margaret Hospital, Hong Kong
  - Queen Elizabeth Hospital, Hong Kong
  - Queen Mary Hospital, Hong Kong
  - Ruttonjee Hospital / Tang Shiu Kin Hospital, Hong Kong
  - Tseung Kwan O Hospital, Hong Kong
  - Tuen Mun Hospital, Hong Kong
  - Tung Wah Hospital, Hong Kong
  - United Christian Hospital, Hong Kong